CLINICAL TRIAL: NCT03725371
Title: Investigation of Psychophysiological Correlation of Aggression and Response to Aversive Stimuli
Status: Completed | Type: Observational
Sponsor: Yale-NUS College (Other)
Responsible Party: Principal Investigator, Jean Liu, Assistant Professor, Yale-NUS College and Adjunct Assistant Professor, Duke-NUS Graduate Medical School, Institute of Mental Health, Singapore
Other Study IDs: YNC-SASSI-Quanti-1
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Conduct Disorder; ADHD; Oppositional Defiant Disorder
MeSH Terms: conditions — Conduct Disorder; Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention was administered for the purpose of this study. — No intervention was administered for the purpose of this study. Observations were carried out for all participants.

SUMMARY:
This study investigates the psychophysiological correlations of aggression and response to aversive stimuli in a population of 133 children clinically diagnosed with conduct disorder (CD) and/or attention-deficit/hyperactivity disorder (ADHD). Data was gathered about participants' level of aggression through the Reactive-Proactive Aggression Questionnaire (RPQ). The stimuli that were presented to the participants included 1) a loud sound, 2) threatening photographs from the International Affective Picture System (IAPS), and 3) the Trier Social Stress Task (TSST). Participants' psychophysiological features of heart rate and galvanic skin conductance were measured and analyzed in relation to their RPQ scores and clinical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between ages 7 and 16 years
2. Subjects who fulfil all criteria for a DSM-IV diagnosis of ADHD, conduct disorder, or oppositional defiant disorder
3. Subjects with willingness to participate in a randomized, double-blind controlled trial
4. Subjects with complete written, informed parental consent and child assent
5. Subjects with IQ of 70 or more

Exclusion Criteria:

1. Subjects who have IQ in the below 70
2. Subjects who are younger than 7 years old or older than 16 years old
3. Those without written parental consent
4. Those with brain pathology such as serious head injury, epilepsy, etc.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study involves children and adolescents diagnosed with disruptive behaviour disorder (DBD, i.e. conduct disorder or oppositional defiant disorder) or attention deficit / hyperactivity disorder (ADHD, i.e. combined type or ADHD predominantly inattentive type or ADHD predominantly hyperactive-impulsive type).
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Heart Rate | 7 minutes
  For Trier Social Stress Task
Skin Conductance Response | 4 minutes
  For loud sound
Skin Conductance Response | 4 minutes
  For threatening photograph

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fung, Study Director — Institute of Mental Health, Singapore

IPD SHARING:
Plan to Share IPD: No